CLINICAL TRIAL: NCT04332146
Title: The Impacts of Mindfulness-based Intervention on Symptoms and Cognition in Chinese Women With Postnatal Depressive Symptoms - A Randomized Controlled Clinical Trial
Brief Title: Mindfulness-based Intervention for Postnatal Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Jingxia Lin, Research Officer, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW17-431
Record Dates: First submitted 2020-03-02; First posted 2020-04-02 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Postnatal Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based intervention (Experimental)
  Interventions: Behavioral: Mindfulness-based program (MBI-p-R)
- Booklet-based psychoeducation group (Active Comparator)
  Interventions: Behavioral: Booklet-based psychoeducation

INTERVENTIONS:
Behavioral: Mindfulness-based program (MBI-p-R) — The MBI-p-R was developed in line with the model of Mindfulness-based Stress Reducation (MBSR) proposed by Kabat-Zinn. It will be conducted for 1.5 hours for each session, once a week for 8 weeks. There are four key operational components to be included in each session: engagement and introduction, mindfulness practices, daily life application, and consolidation of learning.
  Arms: Mindfulness-based intervention
Behavioral: Booklet-based psychoeducation — The participants in the control group will be provided a booklet at baseline, including general information in handling every day stress by a new mother, as well as a record for their weekly activities. The contents covered a range of topics including work-stress, balanced diet, physical exercise, sleeping quality, bonding with baby and the treatment for depression. The participants will be contacted by phone call and/or whatsapp weekly for a short talk based on the record and content on the booklet. They will also be asked to record their daily life weekly for discussion.
  Arms: Booklet-based psychoeducation group

SUMMARY:
Postnatal psychopathology have adverse impact on both mothers and infants. Few postnatal women with depressive symptoms receive treatment, and pharmacological intervention has not been well accepted due to the medication side-effects. Recently, mindfulness-based interventions were found to be beneficial for symptoms in perinatal and antenatal women with depression. These non-pharmacological interventions require less resources and are more feasible for postnatal women to practice at home. To date, no randomized controlled trial has examined mindfulness-based intervention program as a treatment for women with postnatal depression. The proposed randomized controlled trial aims to examine the effects of an 8-week mindfulness-based intervention program on symptom and cognition for postnatal females with depressive symptoms.

A total of 70 postnatal women with depressive symptoms will be recruited from the psychiatric outpatient clinics in Hong Kong, and will be randomized into two groups: 1) an 8-week mindfulness-based intervention program (n=35); 2) a booklet-based psychoeducation control group (n=35). All participants will be assessed for depression, anxiety, stress, cognition, role functioning, quality of life, sleep quality and mindfulness ability at the baseline, 8 weeks, and 3 months after intervention. The intervention sessions will be held once weekly lasting 90 minutes for 8 weeks.

The investigators primarily hypothesize that participants in the mindfulness-based intervention group will improve depressive symptom after 8 weeks compared with the control group. Secondary, the mindfulness-based intervention will improve anxiety, stress, cognitive functions, sleep quality, quality of life and mindfulness ability.

ELIGIBILITY:
Inclusion Criteria:

* Females aged from 18 and above
* The Edinburgh Postnatal Depression Scale cut-off score of >=9
* At least 6 weeks, and up to one and half years after childbirth
* Cantonese-speaking Chinese

Exclusion Criteria:

* Severe physical illness (myocardial infarction, hypertension, fracture, spinal problems in which yoga may be contraindicated), and seizure disorders.
* Comorbid substance dependence
* Women with psychotic depression, severe eating disorders, actively suicidal or obsessive-compulsive disorders
* Known pregnancy
* A history of bipolar disorder, schizophrenia, brain trauma or organic brain disease, mental retardation, or antisocial personality disorder
* Practice of mindfulness (in forms of Tai Chi, Qi gong or yoga etc.) more than twice a week during the previous three months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Depression at 8 weeks | Change from baseline to 8 weeks
  The Edinburgh Postnatal Depression Scale, total score 0-30, higher scores mean worse outcome.
Change from 8 weeks Depression at 3 months | Change from 8 weeks to 3 months
  The Edinburgh Postnatal Depression Scale, total score 0-30, higher scores mean worse outcome.

SECONDARY OUTCOMES:
Change from Baseline Anxiety at 8 weeks | Change from baseline to 8 weeks
  Depression Anxiety Stress Scale, Anxiety subscore 0-42, higher scores mean worse outcome.
Change from 8 weeks Anxiety at 3 months | Change from 8 weeks to 3 months
  Depression Anxiety Stress Scale, Anxiety subscore 0-42, higher scores mean worse outcome.
Change from Baseline Stress at 8 weeks | Change from baseline to 8 weeks
  Depression Anxiety Stress Scale, Stress subscore 0-42, higher scores mean worse outcome.
Change from 8 weeks Stress at 3 months | Change from 8 weeks to 3 months
  Depression Anxiety Stress Scale, Stress subscore 0-42, higher scores mean worse outcome.
Change from Baseline Executive Function at 8 weeks | Change from baseline to 8 weeks
  Trial Making Test, reaction time is recorded, shorter time means better outcome.
Change from 8 weeks Executive Function at 3 months | Change from 8 weeks to 3 months
  Trial Making Test, reaction time is recorded, shorter time means better outcome.
Change from Baseline Attention at 8 weeks | Change from baseline to 8 weeks
  Letter Cancellation Test, correct rate and time are recorded, higher correct rate and shorter time mean better outcome.
Change from 8 weeks Attention at 3 months | Change from 8 weeks to 3 months
  Letter Cancellation Test, correct rate and time are recorded, higher correct rate and shorter time mean better outcome.
Change from Baseline Working Memory at 8 weeks | Change from baseline to 8 weeks
  Digit-Span Test, minimum 0, maximum 14, higher scores mean better outcome.
Change from 8 weeks Working Memory at 3 months | Change from 8 weeks to 3 months
  Digit-Span Test, minimum 0, maximum 14, higher scores mean better outcome.
Change from Baseline Visual-Motor Coordination at 8 weeks | Change from baseline to 8 weeks
  Digit-Symbol-Coding Test, minimum 0, maximum 133, higher scores mean better outcome.
Change from 8 weeks Visual-Motor Coordination at 3 months | Change from 8 weeks to 3 months
  Digit-Symbol-Coding Test, minimum 0, maximum 133, higher scores mean better outcome.
Change from Baseline Role Functioning at 8 weeks | Change from baseline to 8 weeks
  Role Functioning Scale, minimum 4, maximum 38, higher scores mean better outcome.
Change from 8 weeks Role Functioning at 3 months | Change from 8 weeks to 3 months
  Role Functioning Scale, minimum 4, maximum 38, higher scores mean better outcome.
Change from Baseline Quality of Life at 8 weeks | Change from baseline to 8 weeks
  The Short Form Health Survey, minimum score 0, and maximum score 100, higher scores mean better outcome.
Change from 8 weeks Quality of Life at 3 months | Change from 8 weeks to 3 months
  The Short Form Health Survey, minimum score 0, and maximum score 100, higher scores mean better outcome.
Change from Baseline Sleep Quality at 8 weeks | Change from baseline to 8 weeks
  Pittsburg Sleep Quality Index, minimum 0, maximum 21, higher scores mean worse outcome.
Change from 8 weeks Sleep Quality at 3 months | Change from 8 weeks to 3 months
  Pittsburg Sleep Quality Index, minimum 0, maximum 21, higher scores mean worse outcome.
Change from Baseline Mindfulness Levels at 8 weeks | Change from baseline to 8 weeks
  The Five Facet Mindfulness Questionnaire-Revised, minimum 39, maximum 195, higher scores mean better outcome.
Change from 8 weeks Mindfulness Levels at 3 months | Change from 8 weeks to 3 months
  The Five Facet Mindfulness Questionnaire-Revised, minimum 39, maximum 195, higher scores mean better outcome.

OTHER OUTCOMES:
Total attendant classes during the 8-week interventions | At 8 weeks
  The number of classes the participants attended during the 8-week period will be recorded
Self-practice time | At 8 weeks
  How much time the participants spend for self-practice at home will be recorded
Self-practice time | At 3 months
  How much time the participants spend for self-practice at home will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jingxia Lin, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan and clinical study report will be shared through email.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within one year after the completion of the study.